CLINICAL TRIAL: NCT04601662
Title: Evaluation of Corticision-Based Acceleration of Lower Anterior Teeth Alignment on Root Resorption and Dehiscence Formation Using CBCT
Brief Title: Evaluation of the Root Resorption and Dehiscence Formation Between Two Methods of Leveling and Alignment of Lower Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Ortho-06-2020
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticision (Experimental): Patients in this group will be subjected to corticision to accelerate orthodontic movement
  Interventions: Procedure: Corticision
- Traditional treatment (Active Comparator): Patients in this group will undergo normal traditional treatment without any acceleration method.
  Interventions: Other: Traditional Non-accelerated Treatment

INTERVENTIONS:
Procedure: Corticision — A special instrument will be used to cut the cortex of the alveolar bone at different locations between the lower anterior teeth
  Arms: Corticision
Other: Traditional Non-accelerated Treatment — The normal sequence of treatment steps will be followed in this group without using any kind of acceleration methods
  Arms: Traditional treatment

SUMMARY:
The duration of orthodontic treatment is one of the exacerbation causes of orthodontic pain. Several methods have been suggested to reduce the duration of orthodontic treatment classified to surgical and non-surgical methods.

Researchers used minimally invasive surgical methods like corticision, piezocision, micro-osteoperforation, and piezopuncture indicated that most of these methods can accelerate dental movement by 20 - 40%.

The effect of corticision as a minimally invasive procedure on root resorption and dehiscence formation during orthodontic tooth movement has not been studied yet.

Applying corticision on the lower anterior teeth using a surgical blade and a hammer may accelerate tooth alignment during orthodontic treatment. This study consists of two groups, patients will be randomly assigned to one of these two groups.

DETAILED DESCRIPTION:
Orthodontically induced external root resorption accompanying orthodontic treatment is defined as a microscopic loss of root tissue as a result of the inflammatory reaction that occurs in the area of application of orthodontic force. It can be diagnosed and measured using conventional radiography or cone-beam computed tomography (CBCT).

Dehiscence is a loss of alveolar bone on the facial (rarely lingual) aspect of a tooth that leaves a characteristic v-shaped, root-exposed defect from the cementoenamel junction apically. Bone dehiscence cannot be detected through conventional radiography or clinical examination. Actually, CBCT can be considered the best accessible technique providing 3D data.

Corticision is one of the minimally invasive surgical procedures that is not associated with flap lifting. It was used to accelerate tooth movement in animals and case report studies. Its application on humans may aggravate their fear and anxiety towards the pain that may accompany this technique.

No randomized controlled trial (RCT) has compared flapless corticision in the non-extraction-based orthodontic decrowding of lower anterior teeth (LAT) with the conventional treatment in terms of external apical root resorption (EARR) and dehiscence formation (DF).

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 24 years
2. Completion permanent dentition (except third molars)
3. Mild to moderate crowding (2-6 mm according to Little's index)
4. Absence of medications intake that interferes with pain perception for at least one week before the beginning of the treatment

Exclusion Criteria:

1. Medical conditions that would affect tooth movement.
2. Cases which contraindication to oral surgery.
3. Previous orthodontic treatments.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Root Length | T1: one day before the beginning of the orthodontic treatment, T2: exactly at 12 months following the onset of orthodontic treatment
  Cone-beam computed tomography imaging will be used for the lower jaw. Root length will be measured for each root of the six lower anterior teeth The change will be calculated between 'before' and 'after' images in mm.

SECONDARY OUTCOMES:
Change in Dehiscence Proportion | T1: one day before the beginning of the orthodontic treatment, T2: exactly at 12 months following the onset of orthodontic treatment
  Cone-beam computed tomography imaging will be used for the lower jaw. Any V-shaped bone defect located buccally or lingually in the lower anterior region involving bone margin is preliminarily identified as dehiscence. This is going to be measured and the proportion of the presence of such defects will be calculated on two different occasions (T1 and T2).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Radwan Sirri, DDS MSc, Principal Investigator — PhD student, Orthodontics Department, University of Damascus Dental School; Ahmad S Burhan, DDS MSc PhD, Study Director — Professor of Orthodontics, University of Damascus, Damascus, Syria; Fehmieh R Nawaya, DDS MSc PhD, Study Director — Associate Professor of Pedodontics, Syrian Private University, Damascus, Syria
Locations (1):
- Orthodontic Department, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandelaris GA, Neiva R, Chambrone L. Cone-Beam Computed Tomography and Interdisciplinary Dentofacial Therapy: An American Academy of Periodontology Best Evidence Review Focusing on Risk Assessment of the Dentoalveolar Bone Changes Influenced by Tooth Movement. J Periodontol. 2017 Oct;88(10):960-977. doi: 10.1902/jop.2017.160781. PMID 28967331
- [Background] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491
- [Background] Charavet C, Lambert F, Lecloux G, Le Gall M. [Accelerated orthodontic treatment using corticotomies: what are the minimally invasive alternatives?]. Orthod Fr. 2019 Mar;90(1):5-12. doi: 10.1051/orthodfr/2019002. Epub 2019 Apr 17. French. PMID 30994445
- [Background] Makedonas D, Lund H, Hansen K. Root resorption diagnosed with cone beam computed tomography after 6 months and at the end of orthodontic treatment with fixed appliances. Angle Orthod. 2013 May;83(3):389-93. doi: 10.2319/042012-332.1. Epub 2012 Oct 23. PMID 23092202
- [Background] Samandara A, Papageorgiou SN, Ioannidou-Marathiotou I, Kavvadia-Tsatala S, Papadopoulos MA. Evaluation of orthodontically induced external root resorption following orthodontic treatment using cone beam computed tomography (CBCT): a systematic review and meta-analysis. Eur J Orthod. 2019 Jan 23;41(1):67-79. doi: 10.1093/ejo/cjy027. PMID 29771300